CLINICAL TRIAL: NCT02218671
Title: Clinical Pharmacological Study on Absorption From Mucous Membrane of Oral Cavity of WE 941 OD Tablets
Brief Title: Pharmacological Study on Absorption of WE 941 OD Tablets in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 263.506
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- WE 941 OD under deglutition (Experimental)
  Interventions: Drug: WE 941 OD tablets
- WE 941 OD under non-deglutition (Experimental)
  Interventions: Drug: WE 941 OD tablets

INTERVENTIONS:
Drug: WE 941 OD tablets

SUMMARY:
Evaluation whether Brotizolam is absorbed through the mucous membrane of oral cavity when WE 941 OD tablets are administered in Japanese healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* age 20 - 35 years
* body weight 50 - 80 kg
* Body Mass Index (BMI) +/- 20%

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2000-03; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 17 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero to 24hours (AUC0-24 ) | up to 24 hours post dose
Maximum concentration of the analyte in plasma (Cmax) | up to 24 hours
Cmax ratio for non-deglutition to deglutition | up to 24 hours